CLINICAL TRIAL: NCT04978181
Title: The Prevalence and Associated Factors of Early Neurological Deterioration After Successful Recanalization Treatment in Patients With Acute Ischemic Stroke
Brief Title: The Prevalence and Associated Factors of Early Deterioration After Successful Recanalization in Acute Ischemic Stroke
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Osama Ibrahim Aboelfath Ibrahim, osama ibrahim abo-elfath, Assiut University
Other Study IDs: recanalization deterioration
Record Dates: First submitted 2021-07-16; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Acute Stroke
MeSH Terms: conditions — Stroke | interventions — Tissue Plasminogen Activator; Fibrinolytic Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Alteplase Injection — thrombolytic therapy for acute ischemic stroke in time window
  Other Names: thrombolysis

SUMMARY:
stroke is a leading cause of morbidity and mortality worldwide. More than half (54.5%) of the 56.9 million deaths worldwide in 2106 were due to the top 10 causes.

Ischemic heart disease and stroke are the world's biggest killers, accounting for a combined 15.2 million deaths in 2106. These diseases have remained the leading causes of death globally in the last 15 years.

Recent clinical trials have shown that endo-vascular thrombectomy is an effective and safe recanalization modality for acute ischemic stroke patients .

Meta-analysis results show that endovascular treatment is associated with a high ratio of successful recanalization rate and a low rate of symptomatic hemorrhage .

Approximately 2.2-37.5% of patients with acute ischemic stroke might encounter early neurological deterioration (END).

Definition of END: An increase in NIHSS ≥4 or an increase in Ia of NIHSS ≥1 within 72 h after recanalization treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Ischemic stroke of both sex.
2. More than 08 years.
3. Accepting all study requirements.
4. within time window for thrombolysis or thrombectomy
5. fulfilling criteria for thrombolysis or thrombectomy

Exclusion Criteria:

(A)Absolute Contraindications :

1. Intracerebral hemorrhage history or presence on imaging
2. Time of onset more than 465 hours
3. Blood pressure greater than 085/000 mm Hg
4. Recent severe head trauma or neurosurgical intervention
5. Coagulopathy (INR >067, thrombocytopenia, recent use of heparin or direct oral anticoagulants)
6. Endocarditis (infective)
7. Aortic dissection (B)Potential Contraindications :

1.Seizure at onset 2.Noncompressible arterial puncture 3.Recent surgery 4.Gastrointestinal or genitourinary bleeding 5.Multiple cortical microbleeds (>00) 6. Large intracranial aneurysms or arteriovenous malformations 7.Recent transmural myocardial infarction 8. Small NIHSS with nondisabling stroke symptoms

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admittedto Assiut University Hospitals within time window for thrombolysis or thrombectomy within one year are included
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of early neurological deterioration after successful recanalization treatment in patients with acute ischemic stroke | 1 year
  Prevalence of early neurological deterioration after successful recanalization treatment in patients with acute ischemic stroke
factors of deterioration | 1 year
  factors of deterioration

IPD SHARING:
Plan to Share IPD: Undecided